CLINICAL TRIAL: NCT00922428
Title: PASCOE-Agil HOM-Injektopas in the Treatment of Rheumatic Disorders: A Non-interventional Observational Study.
Brief Title: PASCOE-Agil HOM-Injektopas in the Treatment of Rheumatic Disorders
Acronym: 157
Status: Completed | Type: Observational
Sponsor: Pascoe Pharmazeutische Praeparate GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 157 A 07 PA
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Rheumatic Diseases; Arthralgia; Myalgias/Myopathy; Lumbago
Keywords: rheumatism; arthralgia; myalgia; lumbago; homoeopathy; injection; PASCOE-Agil HOM Injektopas; efficacy; tolerability; acceptance; safety
MeSH Terms: conditions — Rheumatic Diseases; Arthralgia; Myalgia; Muscular Diseases; Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational group: Patients suffering from rheumatic disorders of different types and origins, especially those with arthralgia, myalgia, lumbago, or other diagnoses.

SUMMARY:
The purpose of this observational study is to give an overview of the use of PASCOE-Agil HOM-Injektopas in a 2-4 week treatment of rheumatic disorders.

DETAILED DESCRIPTION:
The purpose of this observational study is to give an overview of the use of PASCOE-Agil HOM-Injektopas in a 2-4 week treatment of rheumatic disorders of different aetiology and localisation, displaying a variety of symptoms.

Efficacy and tolerability of the drug will be assessed. Special regard will be taken to the administration management in relation to the Summary of Product Characteristics (SmPC).

ELIGIBILITY:
Due to the design as an Observational Study no inclusion or exclusion criteria for therapy are named. The included patient group is described under "Cohort / Group".

Observational Criteria (=inclusion criteria for documentation):

* Males and females
* At least 18 years old
* Rheumatic disease with accompanying symptoms, e.g. arthralgia, myalgia, lumbago etc.

Exclusion criteria for documentation:

* younger than 18 years
* no Rheumatic disease with accompanying symptoms, e.g. arthralgia, myalgia, lumbago etc.
* no treatment with PASCOE-Agil HOM-Injektopas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of adult patients suffering from rheumatic diseases and relating symptoms who present themselves in German Primary Care Centers.
Sampling Method: Non-Probability Sample
Enrollment: 1389 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anja Braschoss, MD, Study Director — Pascoe Pharmazeutische Praeparate GmbH

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The observational study was carried out by medically-trained doctors who generally treated patients with rheumatic disorders. By choosing a range of different medical specialties - predominantly orthopaedics, rheumatology, general medicine, sports medicine and family doctors - it was ensured that a broad spectrum of patients was recruited.
Pre-assignment Details: The observational study was carried out between January 2008 and the end of May 2008 by 280 therapists. The non-interventional character of an observational study meant that no exact timeframe for the treatment of patients was specified.
Period: Overall Study
Arm/Group | Observational Group
Started | 1389 (13 patients were completely not analysed, 2 not for demographic or efficacy but for safety)
Completed | 1374 (for 11 participants no gender was given)
Not Completed | 15
Not completed — retrospective/extremely implausible data | 2
Not completed — no medication use or questionable use | 13

BASELINE CHARACTERISTICS:
Arm/Group | Observational Group
Number analyzed (Participants) | 1374
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 791
  >=65 years | 580
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (15.5)
Sex/Gender, Customized [Number; unit: participants] — gender of the patients
  participants
    male | 437
    female | 926
    unknown | 11
Region of Enrollment [Number; unit: participants]
  Germany | 1374

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS)
Description: Efficacy of the drug, measured by a Visual Analog Scale (VAS) Scale ranged from 0(=best, no pain) to 10(worst, intolerable pain) The VAS was filled by the patient.
Time Frame: Beginning (Visit 1) and after 2 (visit 2) + 4 weeks (Visit3)
Population: due to character of an observational study: all patient who had a value, descriptive
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Observational (Visit 1): VAS of the observational group at beginning
- Observational Group (Visit 2): VAS of the observational group at visit 2
- Observational Group (Visit 3): VAS of the observational group at visit 3
Arm/Group | Observational (Visit 1) | Observational Group (Visit 2) | Observational Group (Visit 3)
Number analyzed (Participants) | 1368 | 1341 | 1214
units on a scale | 6.57 (1.75) | 4.23 (2.03) | 2.61 (2.03)

2. Primary Outcome: Tolerability of the Drug
Description: Tolerability assessment of medical personnel End of study could by after 2 (visit 2) or after 4 weeks (Visit3).
  It was measured by a score:
  * very well tolerated (no side effects)
  * moderately tolerated (mild side effects)
  * poorly tolerated (marked side effects)
Time Frame: after end of study
Population: 1374 were full analysed, data of 2 patient were additionally analysed for tolerability
Measure: Number; unit: percentage of participants
Arm/Group | Observational Group
Number analyzed (Participants) | 1376
percentage of participants
  moderately/poorly tolerated | 2.8
  well tolerability | 97.2

3. Secondary Outcome: Acceptance of the Drug
Description: Number of patients with good (patient was satisfied with the treatment, there was nothing to complain about) or poor (patient was not satisfied with the treatment, there were ADRs or other reasons) acceptance.
Time Frame: from enrollment until completion
Population: due to the character of an observational study: descriptive
Measure: Number; unit: percentage of participants
Arm/Group | Observational Group
Number analyzed (Participants) | 1374
percentage of participants
  good acceptance | 90.5
  poor acceptance | 8.7

4. Primary Outcome: Pain at Rest
Description: Number of patient (in %) with an improvement of pain at rest between V1 and V2 / V1 and V3 / V2 and V3 A four-point scale (0=not present, 1=slightly, 2=moderate, 3=severe) was used to record symptom severity before the beginning, during treatment and at the end of the observation period.
Time Frame: Beginning (Visit 1) and after 2 (visit 2) + 4 weeks (Visit3)
Population: due to character of an observational study: descriptive, all patients who had an value
Measure: Number; unit: percentage of participants
Groups:
- Observational Group (V1/V2): Improvement in % between Visit 1 and Visit 2
- Observational Group (V1/V3): Improvement in % between Visit 1 and Visit 3
- Observational Group (V2/V3): Improvement in % between Visit 2 and Visit 3
Arm/Group | Observational Group (V1/V2) | Observational Group (V1/V3) | Observational Group (V2/V3)
Number analyzed (Participants) | 1060 | 958 | 945
percentage of participants | 57.5 | 76.8 | 44.1

5. Primary Outcome: Pain in Movement
Description: Number of patients (in %) with an improvement of pain in movement between V1 and V3 / V1 and V3 / V2 and V3 A four-point scale (0=not present, 1=slightly, 2=moderate, 3=severe) was used to record symptom severity before the beginning, during treatment and at the end of the observation period.
Time Frame: Beginning (Visit 1) and after 2 (visit 2) + 4 weeks (Visit3)
Population: due to character of an observational study: descriptive, all patients who had an value
Measure: Number; unit: percentage of participants
Arm/Group | Observational Group (V1/V2) | Observational Group (V1/V3) | Observational Group (V2/V3)
Number analyzed (Participants) | 1322 | 1201 | 1185
percentage of participants | 67.5 | 80.8 | 50.1

6. Primary Outcome: Pain After Rest
Description: Number of patients (in %) with an improvement of pain after rest between V1 and V3 / V1 and V3 / V2 and V3 A four-point scale (0=not present, 1=slightly, 2=moderate, 3=severe) was used to record symptom severity before the beginning, during treatment and at the end of the observation period.
Time Frame: Beginning (Visit 1) and after 2 (visit 2) + 4 weeks (Visit3)
Population: due to character of an observational study: descriptive, all patients who had an value
Measure: Number; unit: percentage of participants
Arm/Group | Observational Group (V1/V2) | Observational Group (V1/V3) | Observational Group (V2/V3)
Number analyzed (Participants) | 1110 | 1012 | 1002
percentage of participants | 60.2 | 78.6 | 49.8

7. Primary Outcome: Pain on Weight-bearing
Description: Number of patients (in%) with an improvement of pain on weight-bearing between V1 and V3 / V1 and V3 / V2 and V3 A four-point scale (0=not present, 1=slightly, 2=moderate, 3=severe) was used to record symptom severity before the beginning, during treatment and at the end of the observation period.
Time Frame: Beginning (Visit 1) and after 2 (visit 2) + 4 weeks (Visit3)
Population: due to character of an observational study: descriptive, all patients who had an value
Measure: Number; unit: percentage of participants
Arm/Group | Observational Group (V1/V2) | Observational Group (V1/V3) | Observational Group (V2/V3)
Number analyzed (Participants) | 1288 | 1165 | 1151
percentage of participants | 64.1 | 79.1 | 50.4

8. Primary Outcome: Morning Stiffness
Description: Number of patients (in%) with an improvement of morning stiffness between V1 and V3 / V1 and V3 / V2 and V3 A four-point scale (0=not present, 1=slightly, 2=moderate, 3=severe) was used to record symptom severity before the beginning, during treatment and at the end of the observation period.
Time Frame: Beginning (Visit 1) and after 2 (visit 2) + 4 weeks (Visit3)
Population: due to character of an observational study: descriptive, all patients who had an value
Measure: Number; unit: percentage of participants
Arm/Group | Observational Group (V1/V2) | Observational Group (V1/V3) | Observational Group (V2/V3)
Number analyzed (Participants) | 941 | 864 | 853
percentage of participants | 54.4 | 74.5 | 42.9

9. Primary Outcome: Tenderness
Description: Number of patients (in%) with an improvement of tenderness between V1 and V3 / V1 and V3 / V2 and V3 A four-point scale (0=not present, 1=slightly, 2=moderate, 3=severe) was used to record symptom severity before the beginning, during treatment and at the end of the observation period.
Time Frame: Beginning (Visit 1) and after 2 (visit 2) + 4 weeks (Visit3)
Population: due to character of an observational study: descriptive, all patients who had an value
Measure: Number; unit: percentage of participants
Arm/Group | Observational Group (V1/V2) | Observational Group (V1/V3) | Observational Group (V2/V3)
Number analyzed (Participants) | 1155 | 1036 | 1023
percentage of participants | 64.5 | 80.8 | 50.3

10. Primary Outcome: Antalgic Position
Description: Number of patients (in%) with an improvement of antalgic position V1 and V3 / V1 and V3 / V2 and V3 A four-point scale (0=not present, 1=slightly, 2=moderate, 3=severe) was used to record symptom severity before the beginning, during treatment and at the end of the observation period.
Time Frame: Beginning (Visit 1) and after 2 (visit 2) + 4 weeks (Visit3)
Population: due to character of an observational study: descriptive, all patients who had an value
Measure: Number; unit: percentage of participants
Arm/Group | Observational Group (V1/V2) | Observational Group (V1/V3) | Observational Group (V2/V3)
Number analyzed (Participants) | 1042 | 931 | 921
percentage of participants | 61.3 | 79.4 | 43.4

ADVERSE EVENTS:
Time Frame: between January 2008 and the end of May 2008
Arm/Group | Observational Group
Serious Adverse Events (participants affected / at risk) | 0/1376
Other Adverse Events (participants affected / at risk) | 23/1376
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Observational Group (N=1376)
Injection site reaction (Injury, poisoning and procedural complications) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No